CLINICAL TRIAL: NCT05772377
Title: An Exploratory Phase II Clinical Trial of Anlotinib Combined With Concurrent Chemoradiotherapy in the Treatment of Locally Advanced Cervical Cancer
Brief Title: Anlotinib Combined With Concurrent Chemoradiotherapy in the Treatment of Locally Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 123321
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: To Evaluate the Efficacy and Safety of Anlotinib Combined With Concurrent Chemoradiotherapy in the Treatment of Locally Advanced Cervical Cancer
MeSH Terms: interventions — Cisplatin; Carboplatin; Brachytherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib+TP then CCRT+Anlotinib (Experimental): Induction regimen:Anlotinib: 10 mg, po, qd, d1-d14, q3w, 2 consecutive cycles Paclitaxel 175mg/m2 intravenous injection for 3 hours, d1；Cisplatin 75mg/m2, iv, divided into 3 days, q3w;Unable to tolerate, nedaplatin 75mg/m2, iv, d1 can be used instead;21 days as a cycle, a total of 2 cycles;Treatment programs:Anlotinib: 10 mg, po, qd, d1-d14, q3w, 2 consecutive cycles;Cisplatin: 30-35 mg/m2, iv, d1, qw, 5 consecutive cycles;Pelvic external radiation therapy: once a day, 1.8-2 Gy/time, 5 days a week, for 5 consecutive weeks, a total of 45-50 Gy;sequential;High dose rate intracavitary radiotherapy: 6 Gy/time, twice a week, 5 consecutive times, a total of 30 Gy/2.5 weeks, bioequivalent dose of 40 Gy sequential Taxane drugs: including but not limited to paclitaxel, nab-paclitaxel, paclitaxel liposome, etc. The dosage regimen is determined by the investigator;Cisplatin 75mg/m2, iv, divided into 3 days, q3w; Unable to tolerate, nedaplatin 75mg/m2, iv, d1 can be used instead;2 cycles
  Interventions: Drug: Hydrochloride anlotinib; Drug: cis Platinum/carboplatin; Radiation: External beam radiotherapy and brachytherapy

INTERVENTIONS:
Drug: Hydrochloride anlotinib — Hydrochloride anlotinib is a small molecular anti-angiogenesis drug with multiple targets. It will be taken at a starting dose of 10 mg for 14 days. Then participants will rest for 7 days and start a new cycles. At most of 3 cycles will be administrated. If intolerable toxicity happen, dosage of 8mg will be taken.
Drug: cis Platinum/carboplatin — Concurrent chemotherapy with cisplatin at 75mg/m2 during radiotherapy will be the most preferred regimen. For patients who cannot tolerate the toxicity of cisplatin, 75 mg/m2 nedaplatin will be used as an alternative drug.
Radiation: External beam radiotherapy and brachytherapy — Radiation will be given by external beam of 40Gy total dose and 3D-brachytherapy of 30Gy/2.5F. Duration of radiotherapy will be no more than 5 weeks

SUMMARY:
To observe the efficacy and safety of hydrochloride anlotinib combined with concurrent radiochemotherapy for patients with FIGO stage IB3 and IIA2-IVA cervical cancer.

DETAILED DESCRIPTION:
Subjects received "anlotinib + paclitaxel/cisplatin" induction therapy for two cycles, and then received "anlotinib + concurrent chemoradiotherapy, sequential high-dose-rate intracavitary radiotherapy, sequential chemotherapy consolidation therapy" regimen:Induction regimen:Anlotinib: 10 mg, po, qd, d1-d14, q3w, 2 consecutive cycles Paclitaxel 175mg/m2 intravenous injection for 3 hours, d1 Cisplatin 75mg/m2, iv, divided into 3 days, q3w;Unable to tolerate, nedaplatin 75mg/m2, iv, d1 can be used instead;21 days as a cycle, a total of 2 cycles

Treatment programs:

Anlotinib: 10 mg, po, qd, d1-d14, q3w, 2 consecutive cycles；Cisplatin: 30-35 mg/m2, iv, d1, qw, 5 consecutive cycles；Pelvic external radiation therapy: once a day, 1.8-2 Gy/time, 5 days a week, for 5 consecutive weeks, a total of 45-50 Gy sequential；High dose rate intracavitary radiotherapy: 6 Gy/time, twice a week, 5 consecutive times, a total of 30 Gy/2.5 weeks, bioequivalent dose of 40 Gy sequential；Taxane drugs: including but not limited to paclitaxel, nab-paclitaxel, paclitaxel liposome, etc. The dosage regimen is determined by the investigator;Cisplatin 75mg/m2, iv, divided into 3 days, q3w;Unable to tolerate, nedaplatin 75mg/m2, iv, d1 can be used instead;2 cycles.A total of 36 patients will be included and this study will be conducted in the department of radiation and clinical oncology in The First Affiliated Hospital of Nanjing Medical University.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the visit; 2. Age ≥ 18 years old (calculated on the date of signing the informed consent); 3. Patients with cervical cancer confirmed by pathology or histology, including squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma, and small cell neuroendocrine carcinoma; 4. Treatment-naïve patients (have not received local treatment or systemic treatment); 5. Locally advanced patients who plan to receive concurrent chemoradiotherapy, FIGO IB3, IIA2-IVA stage (unable/not suitable for pelvic exenteration); 6. There are measurable lesions defined by RECIST standard v1.1; 7. ECOG score 0-1; 8. Expected survival time ≥ 3 months; 9. For non-lactating patients, the serum or urine pregnancy test was negative within 7 days before the study enrollment; female subjects of childbearing age must agree to use high-efficiency methods of contraception during the study period and within 6 months after the last administration of the study drug; 10. The main organ function is good, and the inspection indicators within 14 days before enrollment meet the following requirements:

  1. Blood routine examination (without blood transfusion within 14 days):

     1. Hemoglobin (HB) ≥ 90 g/L;
     2. Neutrophil count (ANC) ≥ 1.5×109/L;
     3. Platelet count (PLT) ≥ 80×109/L;
  2. Biochemical examination:

     1. Total bilirubin ≤ 1.5×ULN (upper limit of normal value);
     2. Blood alanine aminotransferase (ALT) and blood aspartate aminotransferase (AST) ≤ 2.5×ULN; if there is liver metastasis, ALT and AST ≤ 5×ULN;
     3. Serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance ≥ 60mL/min (Cockcroft-Gault formula);
  3. Blood coagulation function test:

     1. Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN;
     2. Doppler ultrasound evaluation: left ventricular ejection fraction (LVE F) ≥ 50%;

Exclusion Criteria:

* 1. Patients with known hypersensitivity to anti-angiogenic drugs or their excipients; 2. Patients with other malignant tumors (except cured carcinoma in situ of the cervix, papillary thyroid carcinoma, basal cell carcinoma of the skin or squamous cell carcinoma of the skin) currently or within the past 5 years; 3. Received radiotherapy, chemotherapy, surgical treatment (excluding local puncture), molecular targeted therapy, immunotherapy or participated in any other drug clinical research within 4 weeks (28 days) before screening (enrolment) or are receiving other clinical trials Study-treated patients (except patients who were followed up for overall survival in a study); 4. Patients with previous or current central nervous system metastases or leptomeningeal disease. Remarks: If the subject has completed radiotherapy or surgery for CNS metastases > 4 weeks before study enrollment, and the subject's nervous system is stable for ≥ 4 weeks (that is, no new neurological deficits caused by brain metastases are found at the time of screening) , central nervous system imaging examination did not find new lesions, and do not need glucocorticoids/steroids for treatment), you can participate in this study; 5. CTCAE ≥ grade 1 (5.0 standard) unresolved toxic reactions caused by any previous treatment, but excluding hair loss; 6. People with multiple factors that affect oral medication (such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.); 7. Imaging studies show that the tumor has invaded around important blood vessels or the researchers judged that the tumor is very likely to invade important blood vessels during the follow-up study and cause fatal massive hemorrhage; 8. There is third space effusion (such as pleural effusion, ascites, pericardial effusion) that cannot be controlled by drainage or other methods; 9. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), bleeding tendency or receiving thrombolytic or anticoagulant therapy; Note: On the premise that the international normalized ratio (INR) of prothrombin time is ≤1.5, the use of low-dose heparin (daily dosage of 0.6-12,000 U for adults) or low-dose aspirin (daily dosage of ≤ 100 U) is allowed for prophylactic purposes. mg); 10. Patients with any severe and/or uncontrolled disease, including:

  1. Patients with hypertension who cannot be well controlled by a single antihypertensive drug treatment (systolic blood pressure > 150 mmHg, diastolic blood pressure > 90 mmHg);
  2. Those with a history of unstable angina; newly diagnosed with angina within 3 months before screening or myocardial infarction within 6 months before screening; arrhythmia (including QTcF: male ≥ 450 ms) requires long-term use of antiarrhythmics Drugs and New York Heart Association grade ≥ II cardiac insufficiency;
  3. Active or uncontrolled severe infection (≥CTCAE 5.0 grade 2 infection);
  4. Those with a history of immunodeficiency, including those who are HIV positive or suffer from other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
  5. Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
  6. Urine routine prompts urine protein ≥ ++, and confirmed 24-hour urine protein quantity > 1.0g;
  7. Patients who have epileptic seizures and need treatment; 11. Regardless of the severity, patients with any bleeding constitution or medical history; within 4 weeks before enrollment, patients with any bleeding or bleeding events CTCAE ≥ grade 3 (5.0 standard), with unhealed wounds, ulcers or fractures; 12. Patients with excessive arterial/venous thrombosis events before enrollment or within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis and pulmonary embolism; 13. Patients with a clear history of neurological or mental disorders, including epilepsy or dementia; 14. Female patients who are pregnant or breastfeeding, female patients who are fertile and have a positive baseline pregnancy test, or female patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial period; 15. According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study;

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
12 months Recurrence-free Survival Rate | 1 years from enrollment
  Proportion of participants free of tumor recurrence 12 months after enrollment

SECONDARY OUTCOMES:
Tumor marker complete response rate | 1 years from enrollment
  Proportion of patients whose CA125, CA199, SCCA, and CEA all fell to the normal range
Progression-free Survival | 2 years from enrollment
  Median time of all participants from enrollment to tumor progression
Objective Response Rate | 2 years from enrollment
  Proportion of participants with complete response and partial response
Overall Survival | 2 years from enrollment
  Median survival time of all participants from enrollment to death of any reason
Adverse events | 2 years from enrollment
  Adverse events data according to CTCAE version 5.0

IPD SHARING:
Plan to Share IPD: No